CLINICAL TRIAL: NCT07307833
Title: Impact of Immunotherapy on Vestibular Function, The Mayo Clinic Arizona Experience
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: MC250709; NCI-2025-08558 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-009510 (Other: Mayo Clinic Institutional Review Board); MC250709 (Other: Mayo Clinic)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphatic System Neoplasm; Malignant Solid Neoplasm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo vestibular function testing with video head impulse testing, sinusoidal harmonic acceleration testing, and pure tone audiometry and complete questionnaires throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study evaluates the impact of immunotherapy on balance in patients receiving immunotherapy as part of their standard of care.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at screening
* Patients who will be initiating single agent immunotherapy with pembrolizumab, cemiplimab, nivolumab, atezolizumab, or dual therapy with (Ipilimumab/Nivolumab or Nivolumab/Relatlimab)

Exclusion Criteria:

* Concurrent chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will be initiating single agent immunotherapy with pembrolizumab, cemiplimab, nivolumab, atezolizumab, or dual therapy with ipilimumab/nivolumab or nivolumab/relatlimab.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2029-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in clinically significant vestibulopathy - vestibular function | Baseline, 3 months, 6 months, 12 months
  Assessed using standard vestibular function testing. Results will be aggregated to determine overall vestibular function. Results from baseline (prior to initiating immunotherapy) will be compared to results at 3, 6, and 12 months.
Change in clinically significant vestibulopathy - hearing level | Baseline,12 months
  Assessed using Pure Tone Audiometry, a standard hearing test. Any change from baseline (prior to initiating immunotherapy) to 12 months will be reported.
Oscillopsia Severity Questionnaire (OSQ) | Baseline, 3 months, 6 months, 12 months
  The OSQ consists of 9 questions to assess visual environment sensation (episodes of oscillopsia). Questions are answered on a 5-point scale: always, often, sometimes, seldom, never. The OSQ is scored by calculating a mean item score, which results in a total score ranging from 1 to 5. A score of 3 or higher indicates moderate to extreme oscillopsia severity.

CONTACTS AND LOCATIONS:
Overall Officials: Carrlene B. Donald, PA-C, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials